CLINICAL TRIAL: NCT03498911
Title: Comparison of Envelope Coronally Advanced Flap and Modified Tunnel Technique in Soft Tissue Dehiscence Coverage Around Implants: A Randomized Clinical Trial
Brief Title: Comparison of Envelope Coronally Advanced Flap and Modified Tunnel Technique in Soft Tissue Dehiscence Around Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Collegiate Professor of Periodontics and Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00140205
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Dental Implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- envelope Coronally Advanced Flap (eCAF) (Active Comparator): A mucogingival surgery where an envelope flap is coronally advanced and sutured to cover the mucosal recession
  Interventions: Procedure: Mucogingival surgery
- Modified Tunnel Technique (MTT) (Experimental): A mucogingival surgery where the gingiva is released without reflecting a flap (as described for tunnel techniques) and then coronally advanced and sutured to cover the mucosal recession
  Interventions: Procedure: Mucogingival surgery

INTERVENTIONS:
Procedure: Mucogingival surgery — The gingiva around the mucosal recession at implant site will be coronally positioned by releasing the underlying mucosa

SUMMARY:
The purpose of this study is to assess the influence of two different flap designs (envelope Coronally Advanced Flap (eCAF) and Modified Tunnel Technique (MTT)) with the addition of a connective tissue graft (CTG) in treating soft tissue dehiscences at implant sites

DETAILED DESCRIPTION:
The primary aim is to compare the test and control groups in terms of:

1. mean mid-facial recession coverage (mRC) measured as a percentage
2. the keratinized tissue (KT) gain measured in mm
3. the keratinized tissue thickness (KTT) gain measured in mm.

The secondary aims are to compare the two groups in terms of:

1. Esthetic score, using numeric values from 0 to 10
2. patient-reported esthetics, using numeric values from 1 to 5
3. patient-reported post-operative pain, based on Visual Analog Scale (VAS) scale, measured as numbers from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Periodontally and systemically healthy
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth)
* Correct implant 3-dimensional position or buccal position ≤ 1 mm
* Buccal soft tissue dehiscence ≤ 4 mm
* Only osseointegrated implants
* The patient must be able to perform good oral hygiene

Exclusion Criteria:

* Contraindications for periodontal surgery
* Patients pregnant or attempting to get pregnant
* Malpositioned implant
* Soft tissue dehiscence (STD) > 4 mm
* Multiple adjacent implants with STD
* Existing of peri-implantitis
* Severe bone loss (≥4mm)
* Moderate-severe interproximal bone loss (implant fixture level to the alveolar bone > 3 mm)
* Moderate-severe papilla height loss (Nordland and Tarnow implant papillae index >1)
* Previous mucogingival surgery around the implant within the past six months or implant placement at the surgical site less than six months prior
* Smoking more than 10 cigarettes a day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
mean mid-facial recession coverage (mRC) | up to 1 year
  mRC measured as a percentage

SECONDARY OUTCOMES:
Esthetic score | 6 months and 1 year
  Esthetic score measured using numeric values from 0 to 10
Patient-reported esthetics | 6 months and 1 year
  Patient-reported esthetics measured using numeric values from 1 to 5
Patient-reported post-operative pain | 2 weeks
  Patient-reported post-operative pain, based on VAS scale, measured as numbers from 0 to 10.
Keratinized tissue (KT) gain | 6 months and 1 year
  KT gain measured in mm
Keratinized tissue thickness (KTT) | 6 months and 1 year
  KTT gain measured in mm

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zucchelli G, Mazzotti C, Mounssif I, Mele M, Stefanini M, Montebugnoli L. A novel surgical-prosthetic approach for soft tissue dehiscence coverage around single implant. Clin Oral Implants Res. 2013 Sep;24(9):957-62. doi: 10.1111/clr.12003. Epub 2012 Aug 27. PMID 22924841
- [Result] Sculean A, Chappuis V, Cosgarea R. Coverage of mucosal recessions at dental implants. Periodontol 2000. 2017 Feb;73(1):134-140. doi: 10.1111/prd.12178. PMID 28000282
- [Result] Schwarz F, Mihatovic I, Shirakata Y, Becker J, Bosshardt D, Sculean A. Treatment of soft tissue recessions at titanium implants using a resorbable collagen matrix: a pilot study. Clin Oral Implants Res. 2014 Jan;25(1):110-5. doi: 10.1111/clr.12042. Epub 2012 Oct 31. PMID 23113567
- [Result] Roccuzzo M, Gaudioso L, Bunino M, Dalmasso P. Surgical treatment of buccal soft tissue recessions around single implants: 1-year results from a prospective pilot study. Clin Oral Implants Res. 2014 Jun;25(6):641-6. doi: 10.1111/clr.12149. Epub 2013 Apr 15. PMID 23582029
- [Result] Morelli T, Neiva R, Nevins ML, McGuire MK, Scheyer ET, Oh TJ, Braun TM, Nor JE, Bates D, Giannobile WV. Angiogenic biomarkers and healing of living cellular constructs. J Dent Res. 2011 Apr;90(4):456-62. doi: 10.1177/0022034510389334. Epub 2011 Jan 19. PMID 21248359
- [Result] Burkhardt R, Joss A, Lang NP. Soft tissue dehiscence coverage around endosseous implants: a prospective cohort study. Clin Oral Implants Res. 2008 May;19(5):451-7. doi: 10.1111/j.1600-0501.2007.01497.x. Epub 2008 Mar 26. PMID 18371102
- [Result] Bassetti RG, Stahli A, Bassetti MA, Sculean A. Soft tissue augmentation around osseointegrated and uncovered dental implants: a systematic review. Clin Oral Investig. 2017 Jan;21(1):53-70. doi: 10.1007/s00784-016-2007-9. Epub 2016 Nov 21. PMID 27873018
- [Result] Anderson LE, Inglehart MR, El-Kholy K, Eber R, Wang HL. Implant associated soft tissue defects in the anterior maxilla: a randomized control trial comparing subepithelial connective tissue graft and acellular dermal matrix allograft. Implant Dent. 2014 Aug;23(4):416-25. doi: 10.1097/ID.0000000000000122. PMID 25033346
- [Derived] Tavelli L, Majzoub J, Kauffmann F, Rodriguez MV, Mancini L, Chan HL, Kripfgans OD, Giannobile WV, Wang HL, Barootchi S. Coronally advanced flap versus tunnel technique for the treatment of peri-implant soft tissue dehiscences with the connective tissue graft: A randomized, controlled clinical trial. J Clin Periodontol. 2023 Jul;50(7):980-995. doi: 10.1111/jcpe.13806. Epub 2023 Apr 4. PMID 36935199